CLINICAL TRIAL: NCT07020858
Title: The Value of FAPI Imaging for the Prediction of Adverse Cardiovascular Events in Chronic Total Occlusion of Coronary Artery Disease (FACT-2 Trial)
Brief Title: FAPI Imaging Predicts Adverse Cardiac Events in Chronic Total Occlusion
Acronym: FACT-2
Status: Recruiting | Type: Observational
Sponsor: Lin Zhao (Other)
Responsible Party: Sponsor-Investigator, Lin Zhao, Cheif of Cardiovascular department, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Other Study IDs: 2025-ke-415
Record Dates: First submitted 2025-06-06; First posted 2025-06-13 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Chronic Total Occlusion (CTO); Chronic Coronary Syndrome
Keywords: Coronary Heart Disease; Major adverse cardiovascular events (MACE); Plaque vulnerability; Optical coherence tomography (OCT); Fibroblast activation protein inhibitor (FAPI); Percutaneous coronary intervention (PCI)
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with at least one untreated CTOat basal angiography: Total occlusion in any major coronary vessel or relevant side branches [reference vessel diameter >2.5 mm or as judged by two independent interventional cardiologists], with TIMI 0 in the distal segment and at least 3 months old
  Interventions: Diagnostic Test: FAPl lmaging

INTERVENTIONS:
Diagnostic Test: FAPl lmaging — Studies have shown that imaging with radionuclide-labeled fibroblast activation protein inhibitor (FAPl) is a reliable technique for detecting myocardial fibrosis and activated CFs in arteries. Preliminary evidence suggests that FAPl imaging can assess plaque characteristics and the status of myocardial fibrosis in various cardiovascular diseases.

SUMMARY:
Prospective, observational, single-center cohort study

Hypothesis Higher myocardial FAPI uptake in CTO patients predicts a greater incidence of major adverse cardiovascular events (MACE) within 12 months after PCI. FAPI PET/CT imaging is associated with plaque vulnerability features and may serve as a non-invasive marker for fibrotic activity and adverse cardiac remodeling.

Inclusion Criteria

* Age ≥ 18 years
* Presence of at least one untreated chronic total occlusion (CTO) lesion in a major coronary artery (diameter ≥ 2.5 mm, TIMI 0 flow for ≥ 3 months) confirmed by coronary angiography or CTCA
* Patient eligible for PCI and undergoing FAPI PET/CT imaging prior to intervention
* Written informed consent provided

Exclusion Criteria

* Allergy or contraindication to antiplatelet agents (aspirin, clopidogrel, or ticagrelor)
* Severe liver dysfunction (liver enzymes >3× upper limit of normal)
* Severe chronic kidney disease (eGFR < 30 mL/min/1.73 m²)
* Estimated life expectancy < 1 year
* Pregnancy or potential for pregnancy

Primary Endpoint Incidence of 1-year MACE, defined as a composite of: Cardiac death, Myocardial infarction, Stroke, Urgent revascularization

Secondary Endpoints

* All-Cause Mortality
* Death from any cause within 12 months
* Quality of Life Change: Measured by Seattle Angina Questionnaire (SAQ): changes in angina frequency, physical limitation, and treatment satisfaction
* Repeat PCI Events: Incidence of: In-stent restenosis (ISR): ≥50% luminal loss in previously stented segment; Target lesion revascularization (TLR): at original PCI lesion; Target vessel revascularization (TVR): other sites in same vessel; De novo lesions: new lesions not previously treated

Sample Size Estimated 470 patients

Follow-Up Duration 12 months post-PCI, One follow-up visit including clinical exam, SAQ questionnaire, imaging (PET/CT, echocardiography), and laboratory testing.

DETAILED DESCRIPTION:
Chronic total occlusion (CTO) of coronary arteries represents one of the most complex and challenging subsets of coronary artery disease and is associated with increased cardiovascular risk. While percutaneous coronary intervention (PCI) for CTO lesions has evolved substantially due to advances in imaging, devices, and operator experience, long-term prognostic evaluation remains suboptimal. In particular, no imaging biomarker currently allows non-invasive prediction of major adverse cardiovascular events (MACE) following CTO PCI.

Fibroblast activation plays a central role in myocardial fibrosis and atherosclerotic plaque instability, both of which contribute to adverse cardiovascular outcomes.

The fibroblast activation protein inhibitor (FAPI), labeled with radionuclides for PET/CT imaging, has recently emerged as a promising tool for quantifying fibrotic activity both in the myocardium and within coronary plaques. Preliminary data from the original FACT study showed that FAPI imaging may predict ventricular remodeling 6 months post-PCI. However, its long-term prognostic value and its role in detecting plaque vulnerability have not been fully evaluated in prospective studies.

The FACT-2 study is a prospective observational cohort study designed to evaluate whether FAPI PET/CT imaging can predict 1-year MACE in patients with CTO undergoing PCI. All enrolled patients will undergo baseline 18F-FAPI PET/CT scans prior to PCI and will be followed for 12 months post-intervention. The study aims to establish a FAPI-based risk stratification model, integrating FAPI uptake parameters with plaque morphology (via OCT and histopathology), serological fibrosis markers, and patient-reported quality of life scores.

The primary endpoint of the study is the incidence of MACE, defined as a composite of cardiac death, myocardial infarction, stroke, and urgent revascularization within one year of PCI. Secondary endpoints include all-cause mortality, repeat PCI events (including in-stent restenosis, target lesion/vessel revascularization, and de novo lesion intervention), and quality of life changes assessed by the Seattle Angina Questionnaire (SAQ).

In this study, FAPI uptake will be quantified by multiple parameters including total uptake volume (FAPI%), standardized uptake values (SUVmax, SUVmean), and target-to-background ratio (TBR). These parameters will be analyzed for correlation with clinical outcomes and histopathological features of plaque vulnerability (e.g., positive remodeling, microcalcification, lipid-rich necrotic core). The goal is to determine whether FAPI PET/CT can serve as a novel imaging biomarker for both myocardial and systemic fibrotic activity and stratify future cardiovascular risk.

By addressing the current evidence gaps in CTO prognosis and risk stratification, the FACT-2 study aims to provide scientific and clinical justification for incorporating molecular imaging into routine management of complex coronary artery disease. This study will also contribute to a more personalized treatment paradigm, bridging the gap between anatomical repair and biologically targeted intervention in cardiovascular medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Confirmed diagnosis of ≥1 untreated chronic total occlusion (CTO):Defined as complete occlusion of a major coronary artery or relevant collateral (reference vessel diameter ≥2.5 mm or confirmed by two independent interventional cardiologists), with TIMI flow grade 0 in the distal segment and duration ≥3 months.Preoperatively confirmed by coronary angiography or coronary computed tomography angiography (CTCA).
3. Willingness to undergo FAPI-PET imaging and receive PCI under imaging guidance.
4. Ability to provide written informed consent.

Exclusion Criteria:

1. Contraindications to antiplatelet therapy: Allergy or intolerance to aspirin, clopidogrel, or ticagrelor.
2. Severe liver dysfunction: Liver function parameters exceeding 3× the upper limit of normal.
3. Severe chronic kidney disease: Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m².
4. Life expectancy <1 year due to non-cardiovascular comorbidities.
5. Pregnancy or women of childbearing potential (unless surgically sterile or using contraception).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with at least one coronary chronic total occlusion (CTO) on coronary angiogram who will be treated by percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 470 (Estimated)
Dates: Start 2025-04-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Major Adverse Cardiovascular Events (MACE) | 12 months after percutaneous coronary intervention (PCI)
  MACE is defined as a composite of cardiac death, myocardial infarction, stroke, and urgent revascularization (including in-stent restenosis, target lesion revascularization, or target vessel revascularization). Events will be assessed through clinical follow-up and hospital record review.

SECONDARY OUTCOMES:
All-Cause Mortality | 12 months post-PCI, verified through national death registry and hospital records.
  Death from any cause, including cardiovascular and non-cardiovascular causes, occurring within 12 months after the index PCI procedure.
Change in Quality of Life | At baseline and 12 months post-PCI.
  Assessed using the Seattle Angina Questionnaire (SAQ). Outcome domains include angina frequency, physical limitation, and treatment satisfaction. Comparison is made between baseline and 12-month follow-up.
Repeat Percutaneous Coronary Intervention (Repeat PCI) | Within 12 months following the index PCI procedure.Angiographic confirmation
  Incidence of repeat PCI due to recurrent or new coronary lesions within 12 months, categorized as:
  In-Stent Restenosis (ISR): ≥50% luminal narrowing in the original stented segment, with or without symptoms.
  Target Lesion Revascularization (TLR): Reintervention at the original stent site due to restenosis or thrombosis.
  Target Vessel Revascularization (TVR): Intervention in the same coronary artery, but outside the original stent site.
  De Novo Lesion: New lesion in a vessel not treated during the index PCI. Confirmation based on follow-up angiography.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Zhao, Dr, Principal Investigator — Beijing Chaoyang Hospital, Capital Medical University, Beijing, China
Locations (1):
- Beijing Chaoyang Hospital，Capital Medical University，Beijing，China, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF
Access Criteria: Need a proposal that describes planned analyses and a data sharing agreement.

REFERENCES:
- [Background] Park TK, Lee SH, Choi KH, Lee JM, Yang JH, Song YB, Hahn JY, Choi JH, Gwon HC, Lee SH, Choi SH. Late Survival Benefit of Percutaneous Coronary Intervention Compared With Medical Therapy in Patients With Coronary Chronic Total Occlusion: A 10-Year Follow-Up Study. J Am Heart Assoc. 2021 Mar 16;10(6):e019022. doi: 10.1161/JAHA.120.019022. Epub 2021 Mar 4. PMID 33660515
- [Background] Werner GS, Hildick-Smith D, Martin Yuste V, Boudou N, Sianos G, Gelev V, Rumoroso JR, Erglis A, Christiansen EH, Escaned J, Di Mario C, Teruel L, Bufe A, Lauer B, Galassi AR, Louvard Y. Three-year outcomes of A Randomized Multicentre Trial Comparing Revascularization and Optimal Medical Therapy for Chronic Total Coronary Occlusions (EuroCTO). EuroIntervention. 2023 Sep 18;19(7):571-579. doi: 10.4244/EIJ-D-23-00312. PMID 37482940
- [Background] Yang L, Guo L, Lv H, Liu X, Zhong L, Ding H, Zhou X, Zhu H, Huang R. Predictors of Adverse Events Among Chronic Total Occlusion Patients Undergoing Successful Percutaneous Coronary Intervention and Medical Therapy. Clin Interv Aging. 2021 Oct 14;16:1847-1855. doi: 10.2147/CIA.S337069. eCollection 2021. PMID 34703218